CLINICAL TRIAL: NCT04830800
Title: A Phase 1/2 Randomized, Placebo-controlled, Observer-blind Trial to Assess the Safety and Immunogenicity of COVIVAC Vaccine Produced by IVAC in Adults Aged 18-60 Years in Vietnam
Brief Title: A Phase 1/2 Safety and Immunogenicity Trial of COVID-19 Vaccine COVIVAC (Phase 1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Vaccines and Medical Biologicals, Vietnam (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVIVAC-0102 (phase 1)
Record Dates: First submitted 2021-03-12; First posted 2021-04-05 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Disease; SARS Pneumonia; Pneumonia, Viral; COVID-19 Vaccine
Keywords: COVID-19; COVIVAC; COVID-19 disease; SARS-CoV-2; COVID-19 vaccine
MeSH Terms: conditions — Pneumonia, Viral; COVID-19 | interventions — COVI-VAC

STUDY DESIGN:
Intervention Model Description: In Phase 1 is dose escalation design, eligible participants will be randomized to received study vaccine or placebo from low dose to higher dose and later to the formulation with CpG adjuvant.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- COVIVAC 1mcg (Experimental): 1mcg IVAC COVIVAC vaccine for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: COVIVAC
- COVIVAC 3mcg (Experimental): 3mcg IVAC COVIVAC vaccine for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: COVIVAC
- COVIVAC 10mcg (Experimental): 10mcg IVAC COVIVAC vaccine for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: COVIVAC
- COVIVAC 1mcg + CpG1018 1.5mg (Experimental): 1mcg + CpG1018 IVAC COVIVAC vaccine for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: COVIVAC
- Placebo (Placebo Comparator): Phosphate buffered saline (pH 7.2) for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: Phosphate-buffered saline

INTERVENTIONS:
Biological: COVIVAC — COVIVAC vaccine, manufactured by IVAC with or without adjuvant CpG1018 for prevention of COVID-19
  Arms: COVIVAC 10mcg; COVIVAC 1mcg; COVIVAC 1mcg + CpG1018 1.5mg; COVIVAC 3mcg
Biological: Phosphate-buffered saline — Phosphate buffer solution (pH 7.2), manufactured by IVAC
  Arms: Placebo

SUMMARY:
This prospective, single-center, randomized, placebo-controlled, observer-blind Phase 1/2 study includes two separate parts.

Part 1 is a first-in-human, Phase 1 study designed to evaluate the safety, tolerability and immunogenicity of the COVIVAC vaccine at three different dose levels (1, 3, and 10 µg) without adjuvant, and at one dose level (1 µg) with the adjuvant CpG 1018, in a total of 120 subjects aged 18-59 years. (Part 2 will be registered in a separate record)

DETAILED DESCRIPTION:
This prospective, single-center, randomized, placebo-controlled, observer-blind Phase 1/2 study includes two separate parts.

Part 1 is a first-in-human, Phase 1 study designed to evaluate the safety, tolerability and immunogenicity of the COVIVAC vaccine at three different dose levels (1, 3, and 10 µg) without adjuvant, and at one dose level (1 µg) with the adjuvant CpG 1018, in a total of 120 subjects aged 18-59 years.

An interim analysis of Phase 1 data conducted after the last subject last visit for V6 (D57) will serve as the basis for decisions about down selection and advancing to Part 2 of the study (Phase 2). Down selection and advancement to Part 2 (Phase 2) will be based on the following parameters:

* Post-dose 2 immunogenicity results at the aggregate treatment level

  o A threshold immune response at Visit 5 (D43) will be required: the observed seroresponse rate in a treatment group (defined as the percentage of subjects with at least a 4-fold rise from baseline in 80% neutralizing antibody titers) will need to be ≥52% at the LL of the 95% CI for that treatment (vaccine formulation) to be considered for advancement to Phase 2.
* Post-dose 1 and post dose 2 safety results including all solicited and unsolicited adverse events, serious adverse events, and clinical laboratory results.

The following process will be followed for the decision about down selection and advancing to Part 2 (Phase 2):

* The DSMB will review the unblinded safety data and provide a recommendation to the Sponsor on whether the safety profile is acceptable for advancing a formulation to Phase 2.
* The Sponsor will review the DSMB recommendation in conjunction with the immunogenicity data and select two formulations to advance to Phase 2.

  o If multiple formulations achieve the threshold immune response (as well as have an adequate safety and tolerability profile per the DSMB), the Sponsor will select two formulations to advance to Phase 2 based on consideration of such factors as the relative functional immunogenicity of these formulations, opportunity for dose sparing, and opportunity to limit cost and possible supply constraints associated with use of the CpG adjuvant.
* The selection and recommendation to advance to Phase 2 along with the interim report will be jointly reviewed by NIHE's IRB and MoH prior to Phase 2 enrollment.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Only:

1. Adult 18 through 59 years of age inclusive at the time of randomization.
2. Healthy, as defined by absence of clinically significant medical condition, either acute or chronic, as determined by medical history, physical examination, screening laboratory test results, and clinical assessment of the investigator.
3. Has provided written informed consent prior to performance of any study-specific procedure.
4. Has a body mass index (BMI) of 17 to 40 kg/m2, inclusive, at screening.
5. Resides in study site area and is able and willing to adhere to all protocol visits and procedures.
6. If a woman is of childbearing potential, must not be breastfeeding or be pregnant (based on a negative urine pregnancy test at screening and during the 24 hours prior to receipt of the first dose of IP), must plan to avoid pregnancy for at least 28 days after the last dose of IP, and be willing to use an adequate method of contraception consistently and have a repeated pregnancy test prior to the second (last) dose of IP.

Exclusion Criteria:

1. Use of any investigational medicinal product within 90 days prior to randomization or planned use of such a product during the period of study participation.
2. History of administration of any non-study vaccine within 28 days prior to administration of study vaccine or planned vaccination within 3 months after enrolment.

   Note: receipt of any COVID-19 vaccine that is licensed or granted Emergency Use Authorization in Vietnam during the course of study participation is not exclusionary if administered after Visit 5.
3. Previous receipt of investigational vaccine for SARS or MERS, or any investigational or licensed vaccine that may have an impact on interpretation of the trial results
4. History of hypersensitivity reaction to any prior vaccination or known hypersensitivity to any component of the study vaccine
5. History of egg or chicken allergy
6. History of angioedema
7. History of anaphylaxis
8. Acute illness (moderate or severe) and/or fever (body temperature measured orally ≥38°C)
9. Any abnormal vital sign deemed clinically relevant by the PI
10. Abnormality in screening laboratory test deemed exclusionary by the PI in consultation with the Sponsor
11. A positive serologic test for hepatitis B (HBsAg) or hepatitis C (HCV Ab)
12. History of confirmed HIV
13. History of laboratory-confirmed COVID-19
14. History of malignancy, excluding non-melanoma skin and cervical carcinoma in situ
15. Any confirmed or suspected immunosuppressive or immunodeficient state
16. Administration of immunoglobulin or any blood product within 90 days prior to first study injection or planned administration during the study period.
17. Administration of any long-acting immune-modifying drugs (e.g., infliximab or rituximab) or the chronic administration (defined as more than 14 days) of immunosuppressants within six months prior to first study injection, or planned administration during the study period (includes systemic corticosteroids at doses equivalent to ≥ 0.5 mg/kg/day of prednisone; the use of topical steroids including inhaled and intranasal steroids is permitted).
18. History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding. (e.g, thalassemia, coagulation factor deficiencies).
19. Recent history (within the past year) or signs of alcohol or substance abuse.
20. Any medical, psychiatric or behavior condition that in the opinion of the PI may interfere with the study objectives, pose a risk to the subject, or prevent the subject from completing the study follow-up.
21. Employee of any person employed by the Sponsor, the contract research organization (CRO), the PI, study site personnel, or site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
There should be an agreement and approval by IRB before sharing IDP

REFERENCES:
- [Derived] Duc Dang A, Dinh Vu T, Hai Vu H, Thanh Ta V, Thi Van Pham A, Thi Ngoc Dang M, Van Le B, Huu Duong T, Van Nguyen D, Lawpoolsri S, Chinwangso P, McLellan JS, Hsieh CL, Garcia-Sastre A, Palese P, Sun W, Martinez JL, Gonzalez-Dominguez I, Slamanig S, Manuel Carreno J, Tcheou J, Krammer F, Raskin A, Minh Vu H, Cong Tran T, Mai Nguyen H, Mercer LD, Raghunandan R, Lal M, White JA, Hjorth R, Innis BL, Scharf R. Safety and immunogenicity of an egg-based inactivated Newcastle disease virus vaccine expressing SARS-CoV-2 spike: Interim results of a randomized, placebo-controlled, phase 1/2 trial in Vietnam. Vaccine. 2022 Jun 9;40(26):3621-3632. doi: 10.1016/j.vaccine.2022.04.078. Epub 2022 May 14. PMID 35577631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The screening and enrollment were conducted from 10 Mar 2021 to 17 April 2021 at the clinical trial center of Hanoi Medical University. Total 224 subjects were screened, and 120 subjects were randomized to 5 treatment arms (25 for each of 4 study vaccine doses/formulation and 20 for placebo cohort).
Pre-assignment Details: This is a first-in-human with dose escalation. There are 4 groups, each group (25 subjects for each vaccine dose/formulation + 5 subject of placebo cohort) will be divided into two sequential subgroups, a sentinel subgroup (n=6) and a larger subgroup (n=24) that includes the remaining subjects to be evaluated at that dose level (or for that formulation in the case of the one adjuvanted treatment group).
Period: Overall Study
Arm/Group | COVIVAC 1mcg | COVIVAC 3mcg | COVIVAC 10mcg | COVIVAC 1mcg + CpG1018 1.5mg | Placebo
Started | 25 | 25 | 25 | 25 | 20
At 14 Days After Second Vaccination | 25 | 25 | 25 | 25 | 20
At Day 197 (6 Months After Second Vaccination) | 23 | 24 | 25 | 24 | 20
Completed | 23 | 24 | 25 | 24 | 20
Not Completed | 2 | 1 | 0 | 1 | 0
Not completed — 4 subject was missing value at visit 7 (Day 197) due to migrated/moved from the study area. | 2 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COVIVAC 1mcg | COVIVAC 3mcg | COVIVAC 10mcg | COVIVAC 1mcg + CpG1018 1.5mg | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 34.4 (11.9) | 36.7 (12.1) | 34.3 (10.6) | 35.1 (11.9) | 32.4 (11.5) | 34.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 12 | 13 | 10 | 58
  Male | 13 | 14 | 13 | 12 | 10 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 25 | 25 | 25 | 25 | 20 | 120
  Kinh (Ethnicity) | 25 | 23 | 25 | 25 | 19 | 117
  Other (Ethnicity) | 00 | 2 | 0 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Vietnam | 25 | 25 | 25 | 25 | 20 | 120
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.1 (2.8) | 22.8 (2.1) | 22.9 (2.5) | 22.3 (2.4) | 22.7 (2.7) | 22.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Solicited Adverse Events
Description: Percentage of participants with solicited local and systemic adverse events (AEs)
Time Frame: During the first 7 days after each vaccination
Population: All participants receiving at least one dose of study vaccine/placebo will be included in the safety analysis population.
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- COVIVAC 1 mcg; COVIVAC 3 mcg; COVIVAC 10 mcg; COVIVAC 1mcg + CpG; Placebo: Participants receiving 2 doses with 28 days apart reporting solicited AEs
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
percent of participants | 88.0 [68.8 to 97.5] | 68.0 [46.5 to 85.1] | 88.0 [68.8 to 97.5] | 80.0 [59.3 to 93.2] | 70.0 [45.7 to 88.1]

2. Primary Outcome: Clinical Safety Tests
Description: Percentage of participants with clinically significant hematological and biochemical abnormalities
Time Frame: At 7 days post each vaccination
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
percent of participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Unsolicited Adverse Events
Description: Number of participants with any unsolicited adverse event
Time Frame: During the first 28 days after each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
percent of participants | 44.0 [24.4 to 65.1] | 32.0 [14.9 to 53.5] | 48.0 [27.8 to 68.7] | 52.0 [31.3 to 72.2] | 45.0 [23.1 to 68.5]

4. Primary Outcome: Serious Adverse Event
Description: Number of participants with serious adverse events (SAEs)
Time Frame: Throughout the Study Period (until Day 197)
Population: There are 116 subject attended the follow-up visit day 197 (23 subjects in 1mcg arm, 24 subjects in 3mcg arm, 25 subjects in 10mcg arm, 24 subjects in 1mcg + CpG arm, and 20 subjects in placebo arm)
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- COVIVAC 1 mcg; COVIVAC 3 mcg; COVIVAC 10 mcg; COVIVAC 1mcg + CpG; Placebo: Participants receiving 2 doses with 28 days apart reporting SAEs
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
percent of participants | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 13.7] | 4.0 [0.1 to 20.4] | 5.0 [0.1 to 24.9]

5. Primary Outcome: Medical Attended Adverse Events
Description: Number of participants with medically-attended AEs (MAAEs)
Time Frame: Throughout the Study Period (until Day 197)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- COVIVAC 1 mcg; COVIVAC 3 mcg; COVIVAC 10 mcg; COVIVAC 1mcg + CpG; Placebo: Participants receiving 2 doses with 28 days apart reporting MAAEs
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
Participants | 3 | 3 | 2 | 2 | 0

6. Primary Outcome: Adverse Event of Special Interest
Description: Number of participants with adverse events of special interest (AESI) , including AESI relevant to COVID-19, and potential immune-mediated medical conditions (PIMMC)
Time Frame: Throughout the Study Period (until Day 197)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- COVIVAC 1 mcg; COVIVAC 3 mcg; COVIVAC 10 mcg; COVIVAC 1mcg + CpG; Placebo: Participants receiving 2 doses with 28 days apart reporting AESIs
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: GMT of 50% Neutralizing Antibody (NT50)
Description: 50% neutralizing antibody (NT50) geometric mean titer (GMT) against SARS-CoV-2 pseudovirus
Time Frame: GMT of NT50 at 28 days after first vaccination, at 14 days and 6 months after the second vaccination
Population: NT50 GMTs are analyzed from subjects with seronegative anti-S IgG at baseline. There were 5 subjects with sero-positive at baseline (anti-S IgG ≥50.3 ELU/mL), 2 subjects (1 μg) with invalid result (IR) at visit 3 (Day 29), 8 subjects missed visit at visit 7 (Day 197), and 1 subject (visit 7 (Day 197)) was not having a sufficient quantity (volume) of specimen to test (QNS- Quantity not sufficient).
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Groups:
- COVIVAC 1 mcg; COVIVAC 3 mcg; COVIVAC 10 mcg; COVIVAC 1mcg + CpG; Placebo: All subjects in the exposed population who have no major protocol deviations that are determined to potentially interfere with the immunogenicity assessment of the study product.
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 24 | 25 | 24 | 25 | 17
IU/ml
  GMT of NT50 at 28 days after first vaccination: number analyzed (Participants) | 22 | 25 | 24 | 25 | 17
  GMT of NT50 at 28 days after first vaccination | 10.67 [6.98 to 16.31] | 8.48 [6.63 to 10.85] | 23.50 [14.91 to 37.02] | 9.35 [6.29 to 13.89] | 5.00 [NA to NA] — All participants in placebo cohort had titer less than 10 and were assigned titer of 5. Then 95%CI had not been calculated for all assigned titers.
  GMT of NT50 at 14 days after second vaccination | 104.96 [69.29 to 159.00] | 170.24 [119.11 to 243.32] | 460.87 [284.49 to 746.58] | 268.32 [175.99 to 409.07] | 5.00 [NA to NA] — All participants in placebo cohort had titer less than 10 and were assigned titer of 5. Then 95%CI had not been calculated for all assigned titers.
  GMT of NT50 at 6 months after second vaccination: number analyzed (Participants) | 21 | 24 | 23 | 22 | 16
  GMT of NT50 at 6 months after second vaccination | 230.72 [75.92 to 701.16] | 607.00 [254.44 to 1448.11] | 556.25 [237.39 to 1303.36] | 452.35 [182.87 to 1118.91] | 20.27 [11.54 to 35.58]

8. Secondary Outcome: Geometric Mean Fold Rise (GMFR)
Description: Geometric mean fold rise (GMFR) (from baseline) in NT50 against SARS-CoV-2 pseudovirus
Time Frame: GMFR at 28 days after first vaccination, at 14 days and 6 months after the second vaccination
Population: There are 2 subjects (1 μg) were invalid result (IR) at visit 3 (Day 29), 8 subjects were missed visit at visit 7 (Day 197), and 1 subject (visit 7 (Day 197)) was not having a sufficient quantity (volume) of specimen to test (QNS- Quantity not sufficient).
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
fold rise
  GMFR at 28 after first vaccination: number analyzed (Participants) | 23 | 25 | 25 | 25 | 20
  GMFR at 28 after first vaccination | 2.06 [1.37 to 3.11] | 1.70 [1.33 to 2.17] | 4.91 [3.15 to 7.66] | 1.87 [1.26 to 2.78] | 1.00 [NA to NA] — All participants in placebo cohort had titer less than 10 and were assigned titer of 5. Then 95%CI had not been calculated for all assigned titers.
  GMFR at 14 days after first vaccination | 22.50 [13.74 to 30.60] | 34.05 [23.82 to 48.66] | 84.75 [51.76 to 138.77] | 53.66 [35.20 to 81.81] | 1.00 [NA to NA] — All participants in placebo cohort had titer less than 10 and were assigned titer of 5. Then 95%CI had not been calculated for all assigned titers.
  GMFR at 6 months after second vaccination: number analyzed (Participants) | 22 | 24 | 24 | 22 | 19
  GMFR at 6 months after second vaccination | 49.53 [17.04 to 143.93] | 121.40 [50.89 to 289.62] | 103.27 [45.14 to 263.28] | 90.47 [36.57 to 223.78] | 4.42 [2.68 to 7.28]

9. Secondary Outcome: Seroresponse in NT50
Description: Percentage of subjects with NT50 seroresponse against SARS-CoV-2 pseudovirus as defined by (1) a ≥ 4-fold increase from baseline, and (2) a ≥ 10-fold increase from baseline
Time Frame: Seroresponse at 28 days after first vaccination, at 14 days and 6 months after the second vaccination
Population: NT50 GMTs are analyzed from subjects with seronegative anti-S IgG at baseline. There were 2 subjects (1 μg) with invalid result (IR) at visit 3 (Day 29), 8 subjects missed visit at visit 7 (Day 197), and 1 subject (visit 7 (Day 197)) was not having a sufficient quantity (volume) of specimen to test (QNS- Quantity not sufficient).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
percentage of participants
  Seroresponse at 28 days after first vaccination: number analyzed (Participants) | 23 | 25 | 25 | 25 | 20
  Seroresponse at 28 days after first vaccination | 13.0 [2.8 to 33.6] | 0.0 [0.0 to 13.7] | 40.0 [21.1 to 61.3] | 8.0 [1.0 to 26.0] | 0.0 [0.0 to 16.8]
  Seroresponse at 14 days after second vaccination | 84.0 [63.9 to 95.5] | 96.0 [79.6 to 99.9] | 96.0 [79.6 to 99.9] | 96.0 [79.6 to 99.9] | 0.0 [0.0 to 16.8]
  Seroresponse at 6 months after second vaccination: number analyzed (Participants) | 22 | 24 | 24 | 22 | 19
  Seroresponse at 6 months after second vaccination | 68.2 [45.1 to 86.1] | 87.5 [67.6 to 97.3] | 87.5 [67.6 to 97.3] | 81.8 [59.7 to 94.8] | 26.3 [9.1 to 51.2]

10. Secondary Outcome: Anti-S IgG GMC
Description: Immunogenicity outcome measurement
Time Frame: GMC of Anti-S IgG at 28 days after the first vaccination, at 14 days and 6 months after the second vaccination
Population: GMCs are analyzed from subjects with seronegative anti-S IgG at baseline. There are 5 subjects were sero-positive at baseline (anti-S IgG ≥50.3 ELU/mL), and 8 subjects were missed visit at visit 7 (Day 197).
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/ml
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
BAU/ml
  GMC of Anti-S IgG at 28 days after first vaccination | 9.89 [6.28 to 15.57] | 15.35 [11.33 to 20.81] | 29.33 [19.26 to 44.66] | 6.40 [4.64 to 8.83] | 3.15 [NA to NA] — All participants had titer below the level of detection. GMCs calculation, concentrations of <10 were assigned as titer of 3.15.
  GMC of Anti-S IgG at 14 days after second vaccination: number analyzed (Participants) | 24 | 25 | 24 | 25 | 17
  GMC of Anti-S IgG at 14 days after second vaccination | 122.54 [87.06 to 172.48] | 173.38 [128.12 to 234.61] | 446.50 [302.60 to 658.83] | 206.51 [152.89 to 278.93] | 3.15 [NA to NA] — All participants had titer below the level of detection. GMCs calculation, concentrations of <10 were assigned as titer of 3.15.
  GMC of Anti-S IgG at 6 months after second vaccination: number analyzed (Participants) | 22 | 24 | 23 | 22 | 16
  GMC of Anti-S IgG at 6 months after second vaccination | 242.54 [129.73 to 909.71] | 469.36 [178.31 to 1235.52] | 515.41 [228.33 to 1163.46] | 350.79 [137.91 to 892.26] | 85.98 [33.22 to 222.51]

11. Secondary Outcome: GMFR in Anti-S IgG GMC
Description: GMFR (from baseline) in anti-S IgG GMC
Time Frame: GMFR at 28 days after the first vaccination, 14 days and 6 months after the second vaccination
Population: There are and 8 subjects were missed visit at visit 7 (Day 197).
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
fold rise
  GMFR at 28 days after first vaccination | 3.00 [1.93 to 4.68] | 4.87 [3.59 to 6.61] | 9.14 [6.10 to 13.69] | 2.03 [1.47 to 2.80] | 1.00 [0.99 to 1.01]
  GMFR at 14 days after second vaccination | 34.65 [23.11 to 51.93] | 55.02 [40.66 to 74.46] | 124.11 [78.20 to 196.99] | 65.54 [48.52 to 88.52] | 0.98 [0.94 to 1.02]
  GMFR at 6 months after second vaccination: number analyzed (Participants) | 23 | 24 | 24 | 22 | 19
  GMFR at 6 months after second vaccination | 103.13 [40.49 to 262.73] | 148.95 [56.59 to 392.10] | 147.60 [65.92 to 330.50] | 111.33 [43.77 to 283.16] | 30.61 [13.60 to 68.88]

12. Secondary Outcome: Seroresponse in Anti-S IgG Concentration
Description: Percentage of subjects with seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline, and (2) a ≥ 10-fold increase from baseline
Time Frame: Seroresponse at 28 days after the first vaccination, 14 days and 6 months after the second vaccination
Population: There are 8 subjects were missed visit at visit 7 (Day 197).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 20
percentage of participants
  Seroresponse at 28 days after first vaccination | 44.2 [35.1 to 53.5] | 44.0 [24.4 to 65.1] | 64.0 [42.5 to 82.0] | 84.0 [63.9 to 95.5] | 0.0 [0.0 to 16.8]
  Seroresponse at 14 days after second vaccination | 82.5 [74.5 to 88.8] | 96.0 [76.9 to 99.9] | 100.0 [86.3 to 100.0] | 100.0 [86.3 to 100.0] | 0.0 [0.0 to 16.8]
  Seroresponse at 6 months after second vaccination: number analyzed (Participants) | 23 | 24 | 24 | 22 | 19
  Seroresponse at 6 months after second vaccination | 82.6 [61.2 to 95.0] | 87.5 [67.6 to 97.3] | 100 [85.8 to 100.0] | 90.9 [70.8 to 98.9] | 89.5 [66.9 to 98.7]

ADVERSE EVENTS:
Time Frame: - Solicited AEs were collected during the 7 days after each vaccination - Unsolicited AEs were collected during the 28 days after each vaccination - MAAEs, AESIs and SAEs were collected from first vaccination until Day 197
Arm/Group | COVIVAC 1 mcg | COVIVAC 3 mcg | COVIVAC 10 mcg | COVIVAC 1mcg + CpG | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 1/25 | 1/20
Other Adverse Events (participants affected / at risk) | 4/25 | 3/25 | 0/25 | 2/25 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVIVAC 1 mcg (N=25) | COVIVAC 3 mcg (N=25) | COVIVAC 10 mcg (N=25) | COVIVAC 1mcg + CpG (N=25) | Placebo (N=20)
Adnexitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COMPLICATED WOUND AT LEFT HAND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVIVAC 1 mcg (N=25) | COVIVAC 3 mcg (N=25) | COVIVAC 10 mcg (N=25) | COVIVAC 1mcg + CpG (N=25) | Placebo (N=20)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT04830800/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT04830800/SAP_001.pdf